CLINICAL TRIAL: NCT04241770
Title: TURKish Acute Myocardial Infarction Registry
Acronym: TURKMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turkish Society of Cardiology (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: TURKMI Study
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Mortality; Registry; Turkey

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
There is no up-to-date information regarding presentation, management and clinical course of patients with acute myocardial infarction (MI) in Turkey. TURKMI registry is designed to provide insight to the characteristics, management from symptom onset to the hospital discharge and outcome of patients with acute MI in Turkey.

DETAILED DESCRIPTION:
Background: There is no up-to-date information regarding presentation, management and clinical course of patients with acute myocardial infarction (MI) in Turkey. TURKMI registry is designed to provide insight to the characteristics, management from symptom onset to the hospital discharge and outcome of patients with acute MI in Turkey.

Methods: TURKMI study, as a nation-wide registry, will be conducted in 50 percutaneous coronary intervention -capable centres selected from each EuroStat NUTS region in Turkey according to their population sampling weight, prioritizing the volume of hospital in each region. All consecutive patients with acute MI admitted to the coronary care units within the 48 hours of symptom onset will be prospectively enrolled during a predefined 2-week period.

The first step of the study has cross-sectional design in which baseline information such as symptoms, risk factors, time periods at each step from symptom onset to revascularization, way of arrival to hospital, biochemical analysis and in-hospital management and outcome will be assessed. The second step has a cohort characteristics in which enrolled patients will be followed-up up to 2 years. Follow-up visits will be conducted at 1st, 6th, 12th and 24th months, and predictors and risk of cardiovascular events, and implementation of guidelines will be assessed as secondary outcomes.

Conclusion: The national TURKMI registry is expected to provide important information to improve the national policy of the diagnosis, management and outcomes of MI in Turkey

ELIGIBILITY:
Inclusion Criteria:

1. having hospitalized within 48 hours of onset of symptoms of the index event
2. had a final (discharge) diagnosis of acute MI either [ST elevation MI (STEMI) or non ST elevation (NSTEMI)] with positive troponin levels, and
3. having signed an Informed Consent. To facilitate consecutive enrolment, all patients hospitalized at each participating site with acute MI will be recruited consecutively during the same 2 consecutive weeks (15 days).

Exclusion Criteria:

1. Patients unwilling or unable to consent will be excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The screened population will consist of all consecutive patients presenting with suspected acute MI in the participating hospitals. Men and women aged ≥18 years will be enrolled if they fulfil the following inclusion criteria;
  1. having hospitalized within 48 hours of onset of symptoms of the index event
  2. had a final (discharge) diagnosis of acute MI either [ST elevation MI (STEMI) or non ST elevation (NSTEMI)] with positive troponin levels, and
  3. having signed an Informed Consent. Patients unwilling or unable to consent will be excluded. To facilitate consecutive enrolment, all patients hospitalized at each participating site with acute MI will be recruited consecutively during the same 2 consecutive weeks (15 days).
Sampling Method: Probability Sample
Enrollment: 1930 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants died | from enrollment till to 2 years follow up
  all cause of death including cardiovascular death

SECONDARY OUTCOMES:
Number of participants developed cardiovascular morbidity | from enrollment till to 2 years follow up
  non-fatal MI, stroke, coronary or peripheral revascularization, emergency department visit due to chest pain or dyspnea, hospitalization for heart failure will be assessed at 1st month and then at every 6 month intervals until the second year.

CONTACTS AND LOCATIONS:
Overall Officials: MUSTAFA K EROL, prof, Study Director — Istanbul Private Sisli International Kolan Hospital,; MERAL KAYIKCIOGLU, prof, Principal Investigator — Ege University School of Medicine Department of Cardiology; MUSTAFa KILICKAP, prof, Principal Investigator — ANKARA University School of Medicine Department of Cardiology
Locations (1):
- Meral Kayikcioglu, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No